CLINICAL TRIAL: NCT00750776
Title: KvaliMed - a Quality Project With Focus on Patients in Antipsychotic Treatment
Acronym: KvaliMed
Status: Terminated | Type: Observational
Why Stopped: Due to lack of financial support
Sponsor: Psychiatric Centre Rigshospitalet (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Anders Fink-Jensen, MD, DMSci, Professor, senior consultant, DMSci, Psychiatric Centre Rigshospitalet
Other Study IDs: NIS-NDK-DUM-2002/1
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Antipsychotic Treatment; Quality Assurance; Medical Treatment
Keywords: Quality assurance; medical treatment; Patient satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Rating and registration in KMS database of all patients in anti-psychotic treatment with 8 selected items from PANSS, GAF, 21 selected items from UKU, 3 selected items from TSQM. and measurement of compliance. Frequency of use of rating scales per participating health care professional.

ELIGIBILITY:
Inclusion Criteria:

* All patients where a physician has decided to treat the patient with antipsychotics.
* All patients that are treated within the Danish health care system

Exclusion Criteria:

* Patients that are treated in accordance with "Law concerning freedom deprivation and other compulsion in psychiatry
* Patients that are in judicial measure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that are treatet with antipsycotic medicine - by a specialist in psychiatry - the patients can stay at the hospital or receive outpatient treatment
Sampling Method: Non-Probability Sample
Enrollment: 212 (Estimated)
Dates: Start 2003-08; Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
GAF score >= 30 or have an improvement on >= 5 points at the GAF scale | All measures are rated every ½ year at least.GAF: At least 85 % of the rated patients must have a score >= 30 or have an improvement on >= 5 points at the GAF scale

SECONDARY OUTCOMES:
PANSS: Share af patients that have a score >= 3 on each an every of the following items P1, P2, P3, N1, N4, N6, G5, G9 | PANSS: At least 70% of the patients have a score <= 3 on each an every of the following items P1, P2, P3, N1, N4, N6, G5, G9
UKU: Share of patients that have a score <=1 on the selected 21 items from the UKU scale | UKU: At least 75 % of the patients have a score on <=1 on the selected items UKU scale.At least 30 % of the patients are examined for metabolic syndrom.
Compliance: Share of patients have according to the specialists evaluation have taken their antipsychotic medicine according to prescription | Compliance: At least 75% of the patients have according to the specialists evaluation taken their antipsychotic medicine according to prescription
Patient satisfaction:Share of patients that scores in one of the to best categories i all selected 3 items in the TSQM scale. | Patient satisfaction:At least 65 % of the patients scores in one of the to best kategories in all the selected 3 items in the TSQM scale.

CONTACTS AND LOCATIONS:
Overall Officials: Soren Blikenberg, Principal Investigator — Research Centre for Psychiatry Vordingborg; Michael Maagensen, Principal Investigator — Children Psychiatry Holbaek; Karin Byrsting, Principal Investigator — Odense University Hospital Odense C Psychiatric Hospital Slagelse; Marianne Jacoby, Principal Investigator — Outpatient TreatmentCopenhagen K; Peter Christoffersen, Principal Investigator — Psychiatric Hospital Slagelse
Locations (10):
- Denmark (10):
  - Research Site, Slagelse, Dianalund
  - Research Site, Bjerringbro
  - Research Site, Brørup
  - Research Site, Copenhagen
  - Research Site, Esbjerg
  - ResearcH Site, Holbæk
  - Research Site, Hviding
  - Research Site, Næstved
  - Research Site, Thyholm
  - Research Site, Varde